CLINICAL TRIAL: NCT02227290
Title: A Phase 4, Double-Blind, Randomized, Vehicle-Controlled, Multicenter, Parallel Group Evaluation of the Efficacy and Safety of Naftin (Naftifine Hydrochloride) Cream, 2% in Pediatric Subjects With Tinea Corporis
Brief Title: Pediatric Subjects With Tinea Corporis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUS90200_4024_1
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Tinea Corporis
Keywords: Tinea Corporis; Ringworm
MeSH Terms: conditions — Tinea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naftin Cream, 2% (Experimental): Once Daily
  Interventions: Drug: Naftin Cream
- Placebo Cream (Placebo Comparator): Once Daily
  Interventions: Drug: Placebo Cream

INTERVENTIONS:
Drug: Naftin Cream
  Arms: Naftin Cream, 2%
Drug: Placebo Cream
  Arms: Placebo Cream

SUMMARY:
The study is being done to see how well the study cream works when applied once a day to affected area of child (where they have ringworm). The results will be compared to those seen with a placebo cream which has no active ingredient. Safety of the cream will also be measured.

DETAILED DESCRIPTION:
The objectives of this study are to evaluate the safety and efficacy of Naftin (naftifine hydrochloride) Cream, 2% applied once daily for 2 weeks, compared to its vehicle in the treatment of pediatric subjects aged 2 to 17 years and 11 months with positive potassium hydroxide (KOH), positive dermatophyte culture, and clinical signs and symptoms of tinea corporis.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females 2 years of age to 17 years, 11 months, of any race. Females of child bearing potential must have a negative urine pregnancy test.
* Presence of tinea corporis by clinical evidence of a tinea infection of at least moderate erythema, moderate induration, and mild pruritus.
* KOH positive and culture positive baseline skin scrapings obtained form the site with the mose severely affected lesion or a representative site of the overall severity.

Exclusion Criteria:

* Tinea infection of the face, scalp, groin, and/or feet
* A life-threatening condition in the opinion of the investigator (ex. autoimmune deficiency syndrome, cancer, etc) within the last 6 months.
* Subjects with abnormal findings- physical or laboratory- that are considered by the investigator to be clinically important and indicative of conditions that might complicate interpretation of study results
* Subjects with a known hypersensitivity or other contradictions to study medications or their components.
* Subjects who have a recent history or who are currently known to abuse alcohol or drugs.
* Uncontrolled diabetes mellitus.
* Hemodialysis or chronic ambulatory peritoneal dialysis therapy.
* Current diagnosis of immunocompromising conditions.
* Current evidence of compromised skin, atopic or contact dermatitis, eczema, impetigo, lichen planus, pityriasis rosea, pityriasis versicolor, psoriasis, seborrhoeic dermatitis and syphilis.
* Severe dermatophytoses, mucocutaneous candidiasis, or bacterial skin infection
* Patients with tinea corporis who have concurrent dermatophytosis of the scalp, beard or nails.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy | Day 21
  Complete cure defined by negative KOH result and negative dermatophyte culture

SECONDARY OUTCOMES:
Secondary Efficacy | Day 21
  Treatment Effectiveness defined as negative KOH, negative culture, and improved sign and symptoms.

OTHER OUTCOMES:
Clinical Success at Days 14 and 21 | Day 14 and Day 21
  Defined as sign and symptom scores of 0 or 1
Clinical cure at Days 14 and 21 | Days 14 and 21
  Defined as erythema, induration, and pruritus score of 0.
Subject Satisfaction | Days 14 and 21
  Assessment on 5 point scale or category of improvement from baseline.
Complete Cure | Day 14
  Defined as negative mycology and abscence of signs/symptoms.
Treatment of Effectiveness | Day 14
  Defined as negative KOH, negative culture, and signs/symptoms.
Mycology Cure | Day 14
  Defined as negative KOH result and negative dermatophyte culture.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Fleischer, MD, Study Director — Merz North America, Inc.
Locations (19):
- United States (14):
  - Merz Investigative Site#001316, Tucson, Arizona
  - Investigative Site# 0010320, Encino, California
  - Merz Investigative Site#001313, Fremont, California
  - Merz Investigative Site#001301, San Diego, California
  - Merz Investigative Site#001312, Miami, Florida
  - Merz Investigative Site#001311, Miami, Florida
  - Merz Investigative Site #001310, Miramar, Florida
  - Merz Investigative Site#001307, Saint Joseph, Missouri
  - Merz Investigative Site#001309, Omaha, Nebraska
  - Merz Investigative Site#001314, Henderson, Nevada
  - Merz Investigative Site#001126, Raleigh, North Carolina
  - Merz Investigative Site#001293, Winston-Salem, North Carolina
  - Investigative Site# 0010319, Gresham, Oregon
  - Merz Investigative Site#001097, Nashville, Tennessee
- Dominican Republic (2):
  - Merz Investigative Site#180002, San Cristóbal
  - Merz Investigative Site# 180001, Santo Domingo
- Merz Investigative Site#504001, San Pedro Sula, Honduras
- Merz Investigative Site#507001, Panama City, Panama
- Merz Investigative Site#001279, Cidra, Puerto Rico